CLINICAL TRIAL: NCT04758884
Title: Telemedicine in Patients with Type 1 Diabetes Mellitus. Efficacy Study of a Specific Virtual Consultation.
Brief Title: Telemedicine in Patients with Type 1 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSAPG-05
Record Dates: First submitted 2021-01-25; First posted 2021-02-17 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Telemedicine; Metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine group (Experimental): Visits by videoconference in months 0, 1, 2, 3, 4 and 6. Additionally, availability to send intermediate messages with a response from the endocrine in less than 72 hours.
  The videoconference will be held safely through the SocialDiabetes® App. Patients will be provided with a glucometer that transfers the data directly to the App without the patient having to enter it to avoid bias in time and value. Videoconferences will NOT be recorded.
  Patients with CGM will additionally have all their values on the platform that corresponds to their sensor (Libreview® for the Freesyle libre® sensor and Clarity® for the Dexcom G5 sensor).
  Interventions: Other: Telemedicine
- Conventional management group (No Intervention): Initial visit, 3 and 6 months.

INTERVENTIONS:
Other: Telemedicine — Visits by videoconference in months 0, 1, 2, 3, 4 and 6.
  Arms: Telemedicine group

SUMMARY:
Management of patients with type 1 Diabetes Mellitus has been changing rapidly in recent years, due in part to the introduction of new technologies such as Apps that recommend insulin boluses, or the use of continuous blood glucose sensors. This fact also entails a change in the care the investigators provide to these patients, facilitating virtual interaction without the need for the patient to go to the consultation, but having all the information necessary to modify treatment doses. There are no studies that compare the influence on glycemic control of conventional management with respect to virtual visits.

The investigators have proposed a randomized cohort study, with the aim to compared the changes in glycated hemoglobin in a group of patients with DM1 of the reference area of the "Hospital Comarcal de l´Alt Penedès" followed by telemedicine respect to the usual management in presential consultation.

DETAILED DESCRIPTION:
Classic management of patients with type 1 diabetes (T1D) by endocrinologists consisted of carrying out a visit every 3-6 months in which HbA1c, microalbuminuria and a notebook with a variable number of annotated controls had been reviewed. In an accelerated way, the management of T1D has clearly been modified with the irruption of new technologies. Devices such as insulin bolus calculators, continuous glucose sensors, or continuous insulin pumps have been appeared and improved. In last months, continuous glucose monitors (CGM) for patients with T1D have been included in public funding in some cases. This fact is also associated with a considerable increase in the number of patient data, and new parameters to analyzed have appeared, with the same importance as HbA1c. Thus, percentage of time in optimal glycemic range, percentage of time in hypoglycemia, coefficient of variation of glycemia, or the mean glycemia are new parameters that the investigators have now been included in the follow-up.

The handling of such amount of data has mainly two repercussions: on the one hand, if these data are well analyzed it is easier to make changes in the treatment, which can conduce to a better disease management such as an improvement in metabolic control or a reduction in hypoglycemia number events. On the other hand, in routine clinical practice it has been found that the fact that patients have higher number of data raises more doubts about theirs treatment and other aspects of their disease, which motivate a greater number of consultations, usually telephone or unscheduled, generating a greater delay in the consultation, occupying spaces assigned to the emergency room or in time slots assigned to other patients.

In this way, telemedicine could be very useful in T1D management. These new devices allow data to be downloaded on secure digital platforms that make it possible for the doctor to have all the patient's blood glucose data without the presential visit of patient to hospital. Some of these platforms also allow safe communication channels between doctors and patients (teleconference, chats). The main benefit that telemedicine can provide is that allow doctors have a very narrow control, unacceptable in routine practice, which allows to interpreted the large volume of data that is generated and to do treatment recommendations, which can improve the metabolic control of the patient.

To date there are few studies on telemedicine in T1D. In this regard, a systematic review reported promising data in terms of HbA1c reduction in 3-6 months interventions, although it do not allow a robust conclusion due to the heterogeneity of the intervention in included studies, the absence of a control group and the small number of patients included2.

Furthermore, the benefits of telemedicine in management of T1D may go beyond the improvement of metabolic control. It must be considered that most T1D patients are young people of working age and that in some areas such as "l´Alt Penedès" there is an important geographical dispersion.

Thus, telemedicine could reduce trips to hospital with benefits on quality of life and reduce indirect costs such as travel costs, lost working hours, etc. In this sense, the Coyote study, carried out in the United States with a sample of 40 T1D subjects between 18-25 years of age, demonstrated that telemedicine was capable of improving the quality of life and saving 6 hours on average between travel to hospital, medical visit and return to work or university1. It should be noted that this study, which is considered a benchmark in its field, did not have a control group nor did it study changes in metabolic control.

On the other hand, being able to establish virtual contact channels between the patient and the doctor with a quick response from the doctor can be reflected in a reduction in the number of unexpected visits or contacts with the Emergency Department. Finally, it must be considered that virtual visits, although they are more frequent than face-to-face ones, are shorter and therefore the total time that doctor spends with the patient does not have to be superior to conventional management.

Hypothesis: Use of telemedicine in patients with T1D allows a closer control of their disease that results in a improve of metabolic control without increasing the number of face-to-face visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1D over 18 years of age
* Duration of T1D greater than 6 months
* Access to smartphones
* In those patients with CGM, the minimum time for handling the sensor before randomization will be 2 months.

Exclusion Criteria:

* Inability to handle smartphones or Apps to manage T1D.
* Admission due to acute decompensation of TD1 in previous 3 months, presence of more than one severe monthly hypoglycemia, or any other circumstance that requires frequent visits and intensive diabetes education
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
To compare changes in HbA1c at 6 months in a group of patients with T1D in the reference area of the "Hospital Comarcal de l´Alt Penedès" followed by telemedicine versus to the usual management in consultation. | 6 months
  HbA1c (%)

SECONDARY OUTCOMES:
Differences in terms of HbA1c at 3 months in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 3 months
  HbA1c at 3 months (%)
Differences in terms of Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL) in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL) (score, minimum value = 43, maximum value = 215, higher scores mean a worse outcome. ).
Differences in terms of episodes of symptomatic hypoglycemia in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Episodes of symptomatic hypoglycemia (number).
Differences in terms of glucometry in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Glucometry: Time in range, above and below range in those patients with CGM (%).
Differences in terms of total time spent by endocrinologist in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Total time spent by endocrinologist (hours).
Differences in terms of indirect costs in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Indirect costs (euros).
Differences in terms of number of unplanned contacts with the specialist in a group of patients with T1D followed by telemedicine versus to the usual management in consultation. | 6 months
  Number of unplanned contacts with the specialist (number).

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Chillarón, Ph.D., Principal Investigator — Consorci Sanitari de l'Alt Penedès
Locations (1):
- Hospital Comarcal de l'Alt Penedès, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballesta S, Chillaron JJ, Inglada Y, Climent E, Llaurado G, Pedro-Botet J, Cots F, Camell H, Flores JA, Benaiges D. Telehealth model versus in-person standard care for persons with type 1 diabetes treated with multiple daily injections: an open-label randomized controlled trial. Front Endocrinol (Lausanne). 2023 Jun 27;14:1176765. doi: 10.3389/fendo.2023.1176765. eCollection 2023. PMID 37441496
- [Background] Raymond JK, Berget CL, Driscoll KA, Ketchum K, Cain C, Fred Thomas JF. CoYoT1 Clinic: Innovative Telemedicine Care Model for Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2016 Jun;18(6):385-90. doi: 10.1089/dia.2015.0425. Epub 2016 May 19. PMID 27196443
- [Background] Peterson A. Improving type 1 diabetes management with mobile tools: a systematic review. J Diabetes Sci Technol. 2014 Jul;8(4):859-64. doi: 10.1177/1932296814529885. Epub 2014 Apr 9. PMID 24876414